CLINICAL TRIAL: NCT05362955
Title: 5-fluorouracil Following Cervical Intraepithelial Neoplasia Treatment Among HIV-positive Women in East Africa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNCPM22120
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: CIN 2/3; HIV Infections
Keywords: cervical cancer; CIN 2/3; 5-Fluorouracil
MeSH Terms: conditions — HIV Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5-FU Arm (Experimental): intravaginal 2g 5-fluorouracil cream in every two weeks
  Interventions: Drug: Intravaginal 5-Fluorouracil (5-FU)

INTERVENTIONS:
Drug: Intravaginal 5-Fluorouracil (5-FU) — Participants will self-administer 2 g of 5% 5-FU intravaginally using an applicator, one night per week (every other week), on weeks 1, 3, 5, 7, 9, 11, 13, 15, for a total of 8 applications.

SUMMARY:
This is a single arm study on the safety, feasibility, and acceptability of adjuvant, self-administered, intravaginal 5-Fluorouracil (5-FU) following treatment for high-grade cervical precancer (CIN2/3) among women living with human immunodeficiency virus (HIV).

ELIGIBILITY:
Subjects must meet all of the inclusion criteria to participate in this study.

Inclusion Criteria:

1. HIV-positive women
2. Age 18 years - 49 years at enrollment
3. Documentation of a biopsy-confirmed CIN2 or CIN3
4. Within 4-12 weeks after primary treatment for CIN2 or CIN3
5. Negative pregnancy test at screening and agreement to use dual form of contraception (hormonal birth control, intrauterine device, or tubal ligation - plus condoms) during the study duration, if of childbearing age.
6. Agree to use dual contraception if of childbearing age (hormonal method, intrauterine or implant device, or tubal ligation - plus condoms) for duration of study
7. Ability to understand and willingness to sign (or assent when applicable) informed consent

Exclusion Criteria:

1. HIV-negative women
2. Pregnant or planning pregnancy within the next 6 months or breastfeeding
3. Unwilling or unable to use birth control during participation in the study
4. History of invasive cervical cancer
5. Untreated vaginal or vulvar dysplasia
6. Known allergy to 5-Fluorouracil
7. History of total hysterectomy
8. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient
9. Current use of chemotherapeutic medication or high dose steroids (10 mg prednisone per day or more (or equivalent steroids)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Safety of intravaginal 5-FU | Up to 5 months
  Safety will be evaluated as type, frequency, and severity of Adverse Events (AE)s. AEs will be evaluated according to the National Institute of Health (NIH) Division of Acquired Immunodeficiency Syndrome (DAIDS) Adverse Event Grading Tables.
  The DAIDS grading table provides an AE severity grading scale ranging from grades 1 to 5. Grade 1 indicates a mild event, Grade 2 indicates a moderate event, Grade 3 indicates a severe event, Grade 4 indicates a potentially life-threatening event and Grade 5 indicates death.

SECONDARY OUTCOMES:
Tolerability of intravaginal 5-FU | Up to 5 months
  Tolerability will be evaluated by assessing the number of participants experiencing specified adverse events (SAEs), defined as a Grade 3 or 4 toxicity that is possibly, probably, or definitely related to the study agent.
Adherence of intravaginal 5-FU | Up to 5 months
  Adherence will be evaluated by assessing the number of participants who are confirmed to use 75% or more of the 5-FU applications.
Acceptability of intravaginal 5-FU | Up to 20 weeks
  Responses to an acceptability questionnaire will be summarized, including means and standard deviation for responses to questions graded on a Likert scale (from 0 to 4), and proportions and 95% confidence intervals for yes/no questions.
Uptake of intravaginal 5-FU | Up to 20 weeks
  The proportion of eligible screened participants who agree to participate in the trial and applied intravaginal 5-FU as the study defined.

CONTACTS AND LOCATIONS:
Overall Officials: Chemtai Mungo, MD, MPH, Principal Investigator — Assistant Professor, Obstetrics and Gynecology
Locations (1):
- Lumumba Sub-County Hospital KEMRI- Research Care Training Program (RCTP) Building, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Adewumi K, Kachoria AG, Adoyo E, Rop M, Owaya A, Tang JH, Rahangdale L, Mungo C. Women's experiences and acceptability of self-administered, home delivered, intravaginal 5-Fluorouracil cream for cervical precancer treatment in Kenya. Front Reprod Health. 2025 Feb 6;7:1487264. doi: 10.3389/frph.2025.1487264. eCollection 2025. PMID 39980670
- [Derived] Adewumi K, Kachoria AG, Adoyo E, Rop M, Owaya A, Tang JH, Rahangdale L, Mungo C. Women's experiences and acceptability of self-administered, home delivered, intravaginal 5-Fluorouracil cream for cervical precancer treatment in Kenya. medRxiv [Preprint]. 2025 Jan 2:2024.08.27.24312651. doi: 10.1101/2024.08.27.24312651. PMID 39568790
- [Derived] Mungo C, Bukusi E, Kirkland GE, Ogollah C, Rota G, Omoto J, Rahangdale L. Feasibility of adjuvant self-administered intravaginal 5-fluorouracil cream following primary treatment of cervical intraepithelial neoplasia grade 2 or 3 among women living with HIV in Kenya: study protocol for a pilot trial. medRxiv [Preprint]. 2023 Dec 14:2023.12.13.23299916. doi: 10.1101/2023.12.13.23299916. PMID 38168442
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials